CLINICAL TRIAL: NCT07335575
Title: Study of Good Clinical Practice Regarding the Use of Physical Restraints in the Emergency Departments of Strasbourg University Hospital
Acronym: PR
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9687
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Physical Restraint
Keywords: Physical Restraint; Emergency departments; Patient safety
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Physical restraint in healthcare settings is an ethical issue. The question of deprivation of liberty, as posed by this practice, has persisted throughout history. In psychiatric wards, physical restraint is governed by strict regulations, enshrined in the Public Health Code. This legal framework is absent from the investigator's emergency departments, despite their frequent involvement in the use of restraint. Several studies have highlighted risk factors associated with restraint. These studies have also highlighted the risks associated with restraint. A best practice guideline published by the French Society of Emergency Medicine (SFMU) in 2021 has provided guidelines for practices within our emergency departments. The objective of this study is to determine whether this guideline is followed by practitioners in the emergency departments of Strasbourg University Hospital. The investigators will also analyze the difference between cases that comply with the recommendations and those that do not. Analyses will also be conducted on the subjects most at risk of restraint, the experiences of restrained patients, the times of day when physical restraint is most likely to be applied, the reasons for restraint, and the nature of the physical and chemical restraint.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18 years)
* Patient who was restrained during their visit to the University Hospital's emergency department between January 1, 2023, and June 30, 2023.

Exclusion Criteria:

Subject (and/or their legal representative, if applicable) must have expressed their objection to the reuse of their data for scientific research purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient (≥18 years) who was restrained during their visit to the University Hospital's emergency department between January 1, 2023, and June 30, 2023.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06-29 (Estimated)

PRIMARY OUTCOMES:
Proportion of cases in accordance with best practice recommendations (in %) | Up to 6 months
  Proportion of cases in accordance with the best practice guidelines of the French Society of Emergency Medicine (SFMU) among all patient cases that underwent physical restraint in the emergency department of the University Hospital over a 6-month period

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Urgences Médico-Chirurgicales Adules - CHU de Strasbourg - France, Strasbourg, France